CLINICAL TRIAL: NCT01011595
Title: Minimally Invasive, Trans-Luminal Diagnosis and Staging of Lung Cancer: A Prospective Head-to-Head Comparison With Traditional Gold Standard Diagnostic Techniques
Brief Title: Minimally Invasive, Diagnosis and Staging of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Society of University Surgeons (Other); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE 09.107
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer
Keywords: lung cancer; mediastinoscopy; mediastinal lymph nodes; staging; EBUS; EUS; Endobronchial Ultrasound; Endoscopic Ultrasound
MeSH Terms: conditions — Lung Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cervical Mediastinoscopy — Surgical Meciastinal Lymph Node Staging
  Other Names: conventional staging procedure
Procedure: Endobronchial Ultrasound (EBUS) — Minimally Invasive Echo-Bronchoscopic Lymph Node Evaluation and Biopsy
  Other Names: Minimally invasive mediastinal staging
Procedure: Endoscopic Ultrasound (EUS) — Minimally Invasive Echo-Endoscopic Lymph Node Evaluation and Biopsy
  Other Names: Minimally invasive mediastinal staging

SUMMARY:
The gold standard techniques to assess the extent of disease and decide on therapy for patients with lung cancer consists of cervical mediastinoscopy, which is a surgical procedure which entails an incision in the neck and the removal of lymph nodes from around the airway. Endobronchial ultrasound (EBUS) and endoscopic ultrasound (EUS) are new, non-surgical techniques that have been available for the past several years and are proving invaluable in lung cancer evaluation. These techniques are minimally invasive and can be performed without surgery.

To date, there have been no head-to-head studies on the same group of patients using both the old and new techniques. The study will consist of a study which compares traditional staging techniques in lung cancer patients to new, less invasive techniques.

The significance of the proposed project is tremendous. If the new strategies prove to be equivalent (or superior) to traditional techniques, these techniques will be considered the new gold-standard tests. This will change the way lung cancer is evaluated. An equivalent or superior result will also significantly impact on patient care, cost and morbidity due to the speed, convenience and lack of operating room requirement as well as the lack of general anesthesia.

DETAILED DESCRIPTION:
1. Problem:

   The gold standard techniques to stage and diagnose the mediastinum in patients with lung cancer consist of cervical mediastinoscopy (CM). CT, PET and PET-CT scans have improved the radiological staging of the mediastinum; however these techniques are unable to provide a tissue diagnosis and are inaccurate. Endobronchial ultrasound (EBUS) and endoscopic ultrasound (EUS) have been available for the past few years and are proving invaluable in the diagnosis and staging of the mediastinum. These techniques rely on imaging of mediastinal lymph nodes (LN) through the airway (EBUS) and the esophagus (EUS) using miniaturized ultrasound probes mounted on the tip of flexible bronchoscopes (EBUS) and esophagoscopes (EUS). Once a LN is visualized and identified using either of these techniques, a needle is passed through the airway (EBUS) or esophageal (EUS) wall into the LN and biopsies are performed. These minimally invasive trans-luminal techniques do not require general anesthesia and can be performed safely, rapidly, accurately and at low cost.

   Due to the cost, inconvenience and risks associated with traditional surgical mediastinal diagnosis and staging, many physicians are foregoing tissue diagnosis of the mediastinum, resulting in incomplete pre-operative staging for patients. The endoscopic techniques are quickly replacing traditional techniques in some centers; however, when replacing a gold standard test with a new modality, one must first prove equivalence in safety and efficacy. Until such a study is completed, we do not have compelling data to be able to offer these techniques as equivalent alternatives to patients. The proposed project will be the first head-to-head comparison of both endobronchial (EBUS) and endoscopic ultrasound (EUS) in addition to transluminal biopsy with gold standard invasive surgical staging techniques in the diagnosis and staging of NSCLC.
2. Objectives:

   * Define and compare the sensitivity, specificity, positive predictive value, negative predictive value, likelihood ratio and accuracies between traditional and minimally invasive mediastinal diagnostic and staging techniques for lung cancer.
   * Compare morbidity, convenience, cost and efficiencies between traditional and minimally invasive diagnostic strategies.
   * Examine the impact on decisions regarding changes in treatment plans (neoadjuvant chemoradiotherapy, prevention of thoracotomy) based on minimally invasive mediastinal staging compared to conventional staging strategies.
3. Methodology:

   The study design consists of a prospective comparison of diagnostic test findings on a consecutive case series with each subject serving as his or her own control. In order to do this, we will enroll N subjects (N=166), and will subject each of the subjects to K procedures (K=3). One of those procedures, the "traditional" one (K-1), is considered to be the gold standard for comparison. We will compare the diagnostic findings from the K-2 and K-3 alternative procedures (EBUS and EUS, respectively) with the gold standard across the N subjects. We will compare them singly and in combination with the gold standard. All patients with a new or suspected diagnosis of lung cancer will be prospectively enrolled in the study. All patients will undergo standard mediastinal staging, EBUS and EUS in the operating room, during one procedure. Patients will be included in the study if they meet one of the following criteria: (A) Lung lesion with mediastinal lymphadenopathy and/or positive PET scan in the mediastinum, (B) Lung lesion without mediastinal lymphadenopathy or positive PET scan in the mediastinum. Sample size has been calculated to be 166 patients.

   Results of traditional staging techniques will be considered as the "gold standard" tests for mediastinal diagnosis and staging. These tests will be used as the standard to which other modalities and combinations of modalities are compared. Data will be collected and analyzed as a whole (all patients with mediastinal LN sampling) and separately based on pre-biopsy diagnosis, post-biopsy diagnosis, mediastinal LN size (CT scan), LN station and PET avidity. Sensitivity, specificity, positive and negative predictive values, likelihood ratios and accuracies will be calculated and used to compare EUS and EBUS (transluminal strategy) to traditional staging, EUS to EBUS, EUS to traditional staging and EBUS to traditional staging. Subanalysis based on pre-biopsy patient and imaging (CT and PET) characteristics as well as ultrasound imaging characteristics during biopsy will be used to develop predictive models for minimally invasive mediastinal diagnosis, in order to better define patients at increased or decreased likelihood of successful diagnosis using these techniques. ROC curves will be constructed and used to discriminate results between diagnostic tests.

   The primary focus of this project and the hypothesis for which the sample size calculations were designed around is whether or not minimally invasive trans-luminal mediastinal LN biopsy is as accurate as traditional "gold standard" techniques in the diagnosis and staging of the mediastinum. Sensitivity, specificity, positive predictive value, negative predictive value and accuracy will be calculated for both strategies (minimally invasive and traditional) and compared. Receiver operating curves will be used to compare the two strategies at differing sensitivity and 1-specificity values. Relative operating characteristic curves will be used to compare the two strategies at different true positive and false positive rates. The study is estimated to be completed in three years. Sample size calculation has determined that 166 patients are required for the study. The thoracic surgery division at the CHUM estimates that accrual will be approximately 1.5 patients per week (6 patients/month).
4. Expected Results:

We expect to find that minimally invasive mediastinal LN staging and diagnosis is not only equivalent in terms of accuracy to traditional staging strategies, but is actually superior. This superiority is possible, secondary to the additional LN basins accessible via these techniques.

ELIGIBILITY:
Inclusion Criteria:

* Lung lesion with mediastinal lymphadenopathy* and/or positive PET scan in the mediastinum
* Lung lesion (>1cm) without mediastinal lymphadenopathy* or positive PET scan in the mediastinum

Exclusion Criteria:

* Age < 18 years old
* CT or PET positivity in an extra-thoracic site (adrenal, liver, brain, bone…)
* Indeterminate pulmonary nodule less than 1cm in diameter without mediastinal lymphadenopathy* on CT and a negative PET scan
* History of previous mediastinoscopy
* Biopsy proven positive mediastinal LN(s)
* Inability to consent for the study
* Cervical or thoracic anatomy precluding mediastinoscopy
* Inability to tolerate general anesthesia
* Pre-operative plan for carinal resection or carinal pneumonectomy (CM contraindicated prior to operative procedure due to additional difficulty secondary to scarring at time of resection)
* Active pulmonary infection (bronchitis, pneumonia)
* Active cutaneous infection overlying proposed surgical site(s)

Lymphadenopathy will be defined as short axis LN diameter of >10 mm on CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the accuracy of the combination of minimally invasive diagnostic tests to correctly diagnose the presence or absence of mediastinal lymph node metastases compared to mediastinoscopy. | 3-6 months
  Define and compare the sensitivity, specificity, positive predictive value, negative predictive value, likelihood ratio and accuriacies between traditional and minimally invasive mediastinal diagnostic and staging techniques for lung cancer.

SECONDARY OUTCOMES:
The safety of all diagnostic techniques will be evaluated and compared between techniques. | 3-6 months
  Compare morbidity, convenience, cost and efficiencies between traditional and minimally invasive diagnostic strategies.
Procedure-related morbidity | 3-6 months
Procedural, hopsitalization and overall cost | termination of enrollment
Clinical decision making realted to diagnostic technique results. | termination of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Liberman M, Sampalis J, Duranceau A, Thiffault V, Hadjeres R, Ferraro P. Endosonographic mediastinal lymph node staging of lung cancer. Chest. 2014 Aug;146(2):389-397. doi: 10.1378/chest.13-2349. PMID 24603902